CLINICAL TRIAL: NCT06771778
Title: Elevating the Neonatal Dietitian for the Future: Insights From the Experts Themselves
Brief Title: Advancing the Role of the Neonatal Registered Dietitian Nutritionist
Status: Completed | Type: Observational
Sponsor: Florida International University (Other)
Collaborators: The Rickard Foundation, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-23-0559
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Opinions of the Neonatal Registered Dietitian
Keywords: Neonatal Intensive Care Unit; Neonatal Dietitian Nutritionist; Neonatal Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn Intensive Care Unit (NICU) Registered Dietitian(s): Current or former Newborn Intensive Care Unit (NICU) Registered Dietitian(s)
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — A Qualtrics link was provided for current and former NICU RDNs to complete a 10-minute online survey that provided an optional gift card for completion. Part 1 of the survey had eight questions, and part 2 had eleven additional questions.

SUMMARY:
This observational study aims to identify the needs, engagement levels, and expertise of NICU RDNs and provide insights into their job satisfaction and career longevity.

This cross-sectional examination was conducted in March - April 2024 using a national, online, IRB-approved survey sent to established Neonatal and Pediatric Dietitian practice groups. A Qualtrics link was provided for current and former NICU RDNs to complete a 10-minute online survey.

ELIGIBILITY:
Inclusion Criteria: Current and former Neonatal Registered Dietitian(s)

-

Exclusion Criteria:

Practice outside of the USA and Canada.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Current and former Neonatal Registered Dietitian.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Exploratory Neonatal Registered Dietitian Opinions | Time Frame: March 28 - April 2, 2024
  Description: 253 current (n=206) and former (n=47) NICU RDNs completed the online questionnaire. Multiple choice, observational data collected.

CONTACTS AND LOCATIONS:
Overall Officials: Alayne M Gatto, M.S., R.D.N., Study Chair — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unsure of current submission time-frame and publication.

REFERENCES:
- [Derived] Abel DM, Gatto AM, Fowler JO, Valentine CJ. Elevating the role and professional contributions of the neonatal dietitian for the future: insights from the experts themselves. Front Pediatr. 2025 Aug 26;13:1639283. doi: 10.3389/fped.2025.1639283. eCollection 2025. PMID 40933702